CLINICAL TRIAL: NCT00004212
Title: A Phase I Dose Escalation Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Pediatric Patients With Advanced Solid Tumors and Lymphomas
Brief Title: DX-8951f in Treating Children With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067330; DAIICHI-8951A-PRT013; MSKCC-99071; UTHSC-9895011445; NCI-V99-1573
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood craniopharyngioma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; childhood central nervous system germ cell tumor; unspecified childhood solid tumor, protocol specific; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood choroid plexus tumor; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; untreated childhood supratentorial primitive neuroectodermal tumor; recurrent childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood medulloblastoma; recurrent childhood medulloblastoma; untreated childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway and hypothalamic glioma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Recurrence; Astrocytoma; Oligodendroglioma; Choroid Plexus Neoplasms; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Optic Nerve Glioma; Familial ependymoma | interventions — Filgrastim; exatecan

INTERVENTIONS:
Biological: filgrastim
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of DX-8951f in treating children who have advanced solid tumors or lymphomas that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of exatecan mesylate (DX-8951f) with and without filgrastim (G-CSF) in pediatric patients with advanced solid tumors or lymphomas.
* Determine the toxic effects, including dose-limiting toxicity, of exatecan mesylate in these patients.
* Determine the pharmacokinetics of exatecan mesylate in these patients.
* Determine the recommended dose of exatecan mesylate for phase II study.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of exatecan mesylate (DX-8951f). Patients are stratified according to prior treatment (minimally treated vs heavily treated).

Patients receive exatecan mesylate IV over 30 minutes daily for 5 days. Patients in dose levels 5 and above also receive filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing for at least 7 days or until blood counts recover. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of exatecan mesylate with and without G-CSF until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumors, including brain tumors and lymphomas, that have failed standard therapy (surgery, radiotherapy, endocrine therapy, or chemotherapy) or for which no standard therapy exists

  * Histology requirement waived for brain stem gliomas

PATIENT CHARACTERISTICS:

Age:

* 21 and under at diagnosis

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 750/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 8.5 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT or SGPT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases)

Renal:

* Creatinine no greater than 1.5 times ULN OR
* GFR at least 70 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No history of severe or life-threatening hypersensitivity to camptothecin analogs
* HIV negative
* No other concurrent severe or uncontrolled medical illness
* No systemic infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior immunotherapy

Chemotherapy:

* See Disease Characteristics
* Recovered from prior chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior extensive radiotherapy involving cranial, whole pelvic, or at least 25% of bone marrow reserve
* Recovered from prior radiotherapy
* Concurrent localized radiotherapy for pain allowed

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* No other concurrent antitumor therapy
* No concurrent drugs that induce or inhibit CYP3A enzyme

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Institute for Drug Development, San Antonio, Texas